CLINICAL TRIAL: NCT01500278
Title: A Multicenter, Single-blind, Randomized Parallel-group Study to Assess the Short- and Long-term Efficacy of Certolizumab Pegol Plus Methotrexate Compared to Adalimumab Plus Methotrexate in Subjects With Moderate to Severe Rheumatoid Arthritis Responding Inadequately to Methotrexate
Brief Title: Study to Assess the Short- and Long-term Efficacy of Certolizumab Pegol Plus Methotrexate Compared to Adalimumab Plus Methotrexate in Subjects With Moderate to Severe Rheumatoid Arthritis (RA) Inadequately Responding to Methotrexate
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: UCB Pharma SA (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RA0077; 2011-002067-20 (EudraCT Number)
Expanded Access: NCT03559686 (Available)
Record Dates: First submitted 2011-12-22; First posted 2011-12-28 (Estimated); Results first posted 2017-03-31 (Actual); Last update posted 2018-07-31 (Actual); Status verified 2017-07

CONDITIONS: Rheumatoid Arthritis
Keywords: Certolizumab Pegol; Cimzia; Adalimumab; Humira; Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Certolizumab Pegol; Adalimumab; Methotrexate

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Certolizumab Pegol + Methotrexate (CZP + MTX) (Active Comparator)
  Interventions: Biological: Certolizumab Pegol (CZP); Drug: Methotrexate (MTX)
- Adalimumab + Methotrexate (ADA + MTX) (Active Comparator)
  Interventions: Biological: Adalimumab (ADA); Drug: Methotrexate (MTX)
- CZP + MTX followed by ADA + MTX (Active Comparator): Those subjects who received Certolizumab Pegol (400 mg at Weeks 0, 2, 4 followed by 200 mg every two weeks) + Methotrexate (CZP+ MTX) at Baseline and are Non-Responders at Week 12, switch to Adalimumab (40 mg) + Methotrexate (ADA + MTX) after Week 12.
  Interventions: Biological: Certolizumab Pegol (CZP); Biological: Adalimumab (ADA); Drug: Methotrexate (MTX)
- ADA + MTX followed by CZP + MTX (Active Comparator): Those subjects who received Adalimumab (40 mg + Placebo at Weeks 0, 2, 4 followed by 40 mg ADA every two weeks) + Methotrexate (ADA+ MTX) at Baseline and are Non-Responders at Week 12, switch to Certolizumab Pegol (400 mg at Weeks 12, 14, 16 followed by 200 mg every two weeks) + Methotrexate (CZP+ MTX) after Week 12.
  Interventions: Biological: Certolizumab Pegol (CZP); Biological: Adalimumab (ADA); Drug: Methotrexate (MTX)

INTERVENTIONS:
Biological: Certolizumab Pegol (CZP) — * Active substance: an injectable volume of 1 ml solution for injection CZP
  * Pharmaceutical form: prefilled syringes CZP
  * Concentration: 200 mg/ml CZP
  * Route of Administration: injections will be given subcutaneously: loading dose of CZP 400 mg at Baseline, and Weeks 2 and 4, followed by a maintenance dose of 200 mg every 2 weeks through Week 102 or withdrawal.
  Other Names: Cimzia; CZP
  Arms: ADA + MTX followed by CZP + MTX; CZP + MTX followed by ADA + MTX; Certolizumab Pegol + Methotrexate (CZP + MTX)
Biological: Adalimumab (ADA) — * Active substance: an injectable volume of 0.8 ml solution for injection ADA
  * Pharmaceutical form: prefilled syringes ADA
  * Concentration: 40 mg/0.8 ml ADA
  * Route of Administration: injections will be given subcutaneously. ADA 40 mg plus an injection with Placebo (to preserve blind) at Baseline, and Weeks 2 and 4, followed by ADA 40 mg every 2 weeks through Week 102 or withdrawal.
  Other Names: Humira; ADA
  Arms: ADA + MTX followed by CZP + MTX; Adalimumab + Methotrexate (ADA + MTX); CZP + MTX followed by ADA + MTX
Drug: Methotrexate (MTX) — * Active substance: Methotrexate
  * Pharmaceutical form: oral tablet
  * Concentration: 15-25 mg/week
  * Route of Administration: MTX orally
  Other Names: MTX

SUMMARY:
This study is conducted to evaluate the short (12 Weeks) and long term (104 Weeks) efficacy of Certolizumab Pegol compared with Adalimumab both in combination with Methotrexate (MTX) in the treatment of moderate to severe Rheumatoid Arthritis (RA) that is not responding adequately to MTX.

ELIGIBILITY:
Inclusion Criteria:

* Subject must have a diagnosis of Rheumatoid Arthritis (RA) at Screening, as defined by the 2010 European League Against Rheumatism (EULAR)/American College of Rheumatology (ACR) classification criteria (Aletaha D et al, 2010)
* Subject must have a positive Rheumatoid Factor (RF) and/or a positive anti-Cyclic Citrullinated Peptide antibody (anti-CCP) as determined by the central laboratory at Screening
* Subject must have moderate to severe RA disease at Screening and Baseline defined as:

  1. Screening (all criteria required)

     * ≥ 4 swollen joints (of 28 prespecified joints)
     * Disease Activity Score [Erythrocyte Sedimentation Rate] (DAS28[ESR]) > 3.2
     * C-Reactive Protein (CRP) concentration ≥ 10 mg/L (or 1.0 mg/dL) or Erythrocyte Sedimentation Rate (ESR) (Westergren) ≥ 28 mm/hr
  2. Baseline (both criteria required)

     * ≥ 4 swollen joints (of 28 prespecified joints)
     * Disease Activity Score [Erythrocyte Sedimentation Rate] (DAS28[ESR]) > 3.2
* Subject must have inadequately responded previously to Methotrexate (MTX)
* Subject is using MTX 15 to 25 mg/week orally or subcutaneously at Screening and has used the same MTX regimen for a minimum of 28 days prior to Baseline

Exclusion Criteria:

* Subject has previously received any biological Disease Modifying Antirheumatic Drug (DMARD) or has received treatment with cyclophosphamide, chlorambucil, Janus Kinase, phosphodiesterase 4 inhibitors or investigational agents such as spleen tyrosine kinase
* Diagnosis of any other inflammatory arthritis
* Infected with Tuberculosis (TB) or high risk of acquiring TB infection
* Subjects with concurrent acute or chronic viral hepatitis B or C infection
* Subjects with a history of chronic or recurrent infections or subjects at high risk of infection
* Use of prohibited medications like nonbiological DMARDs (excluding MTX), biological DMARDs excluding study medications, experimental therapy, IA hyaluronic acid

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 915 (Actual)
Dates: Start 2011-12; Primary Completion 2015-11 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — +1 877 822 9493 (UCB)
Locations (175):
- United States (62):
  - 141, Birmingham, Alabama
  - 214, Tuscaloosa, Alabama
  - 159, Tucson, Arizona
  - 152, Hot Springs, Arkansas
  - 147, Covina, California
  - 161, Fullerton, California
  - 217, La Mesa, California
  - 149, Los Angeles, California
  - 144, Menifee, California
  - 185, Roseville, California
  - 208, Sacramento, California
  - 189, Van Nuys, California
  - 148, Whittier, California
  - 220, Lewes, Delaware
  - 142, Aventura, Florida
  - 216, Fort Lauderdale, Florida
  - 162, Gainesville, Florida
  - 209, Vero Beach, Florida
  - 145, Coeur d'Alene, Idaho
  - 202, Maywood, Illinois
  - 134, Lexington, Kentucky
  - 178, Baltimore, Maryland
  - 137, Battle Creek, Michigan
  - 153, Detroit, Michigan
  - 155, Lansing, Michigan
  - 204, Eagan, Minnesota
  - 180, Rochester, Minnesota
  - 143, Saint Louis Park, Minnesota
  - 135, Omaha, Nebraska
  - 170, Reno, Nevada
  - 201, Teaneck, New Jersey
  - 150, Voorhees Township, New Jersey
  - 205, Albuquerque, New Mexico
  - 154, Albany, New York
  - 136, Brooklyn, New York
  - 219, Orchard Park, New York
  - 207, Plainview, New York
  - 167, Syracuse, New York
  - 140, Cincinnati, Ohio
  - 184, Oklahoma City, Oklahoma
  - 164, Bethlehem, Pennsylvania
  - 132, Duncansville, Pennsylvania
  - 190, Wyomissing, Pennsylvania
  - 210, Charleston, South Carolina
  - 187, Myrtle Beach, South Carolina
  - 203, Orangeburg, South Carolina
  - 133, Jackson, Tennessee
  - 160, Knoxville, Tennessee
  - 138, Austin, Texas
  - 151, Corpus Christi, Texas
  - 131, Dallas, Texas
  - 146, Dallas, Texas
  - 213, Dallas, Texas
  - 166, Houston, Texas
  - 212, Houston, Texas
  - 139, San Antonio, Texas
  - 181, Sugar Land, Texas
  - 165, Victoria, Texas
  - 211, Arlington, Virginia
  - 157, Spokane, Washington
  - 163, Clarksburg, West Virginia
  - 215, Glendale, Wisconsin
- Australia (8):
  - 6, Camperdown, New South Wales
  - 5, Kogarah, New South Wales
  - 2, Maroochydore, Queensland
  - 4, Hobart, Tasmania
  - 7, Clayton, Victoria
  - 8, Fitzroy, Victoria
  - 1, Malvern, Victoria
  - 3, Subiaco, Western Australia
- Austria (2):
  - 85, Stockerau
  - 22, Vienna
- Bulgaria (6):
  - 18, Pleven
  - 35, Plovdiv
  - 21, Sofia
  - 29, Sofia
  - 34, Sofia
  - 46, Sofia
- Canada (13):
  - 179, Edmonton, Alberta
  - 168, St. John's, Newfoundland and Labrador
  - 176, St. John's, Newfoundland and Labrador
  - 183, Halifax, Nova Scotia
  - 172, Hamilton, Ontario
  - 174, Hamilton, Ontario
  - 177, Ottawa, Ontario
  - 206, Ottawa, Ontario
  - 175, St. Catharines, Ontario
  - 218, Rimouski, Quebec
  - 169, Sainte-Foy, Quebec
  - 221, Barrie
  - 171, Québec
- Czechia (5):
  - 103, Brno
  - 61, Hradec Králové
  - 58, Pilsen
  - 49, Prague
  - 40, Uherské Hradiště
- France (6):
  - 89, Brest
  - 70, Le Mans
  - 62, Lyon
  - 72, Montpellier
  - 90, Orléans
  - 105, Toulouse
- Germany (12):
  - 56, Berlin
  - 64, Cologne
  - 47, Fulda
  - 17, Hamburg
  - 31, Heidelberg
  - 37, Herne
  - 63, Osnabrück
  - 11, Ratingen
  - 66, Rheine
  - 48, Rostock
  - 71, Traunstein
  - 44, Zerbst
- Greece (2):
  - 94, Heraklion
  - 95, Larissa
- Hungary (6):
  - 13, Budapest
  - 42, Budapest
  - 68, Gyula
  - 100, Kistarcsa
  - 43, Szeged
  - 33, Veszprém
- Ireland (3):
  - 23, Dublin
  - 51, Dublin
  - 20, Limerick
- Italy (8):
  - 80, Bergamo
  - 38, Genova
  - 88, Genova
  - 79, Magenta
  - 98, Napoli
  - 67, Prato
  - 36, Roma
  - 39, Verona
- Mexico (5):
  - 194, Chihuahua City
  - 195, Chihuahua City
  - 193, Guadalajara
  - 192, Monterrey
  - 191, San Luis Potosí City
- 60, Monaco, Monaco
- Poland (5):
  - 107, Bydgoszcz
  - 106, Poznan
  - 113, Warsaw
  - 115, Warsaw
  - 108, Wroclaw
- Portugal (5):
  - 69, Coimbra
  - 27, Lisbon
  - 76, Lisbon
  - 14, Ponte de Lima
  - 81, Porto
- Romania (10):
  - 54, Bacau
  - 74, Brăila
  - 24, Bucharest
  - 25, Bucharest
  - 28, Bucharest
  - 32, Bucharest
  - 57, Bucharest
  - 12, Cluj-Napoca
  - 96, Galati
  - 26, Iași
- Spain (6):
  - 16, A Coruña
  - 52, A Coruña
  - 30, Madrid
  - 83, Madrid
  - 82, Sabadell
  - 65, Vigo
- Switzerland (2):
  - 53, Sankt Gallen
  - 50, Zurich
- United Kingdom (8):
  - 86, Ashford
  - 78, Brighton
  - 59, Leeds
  - 19, London
  - 77, Poole
  - 55, Sheffield
  - 73, Upton
  - 99, Wigan

REFERENCES:
- [Result] Smolen JS, Burmester GR, Combe B, Curtis JR, Hall S, Haraoui B, van Vollenhoven R, Cioffi C, Ecoffet C, Gervitz L, Ionescu L, Peterson L, Fleischmann R. Head-to-head comparison of certolizumab pegol versus adalimumab in rheumatoid arthritis: 2-year efficacy and safety results from the randomised EXXELERATE study. Lancet. 2016 Dec 3;388(10061):2763-2774. doi: 10.1016/S0140-6736(16)31651-8. Epub 2016 Nov 15. PMID 27863807
- [Derived] Smolen JS, Taylor PC, Tanaka Y, Takeuchi T, Hashimoto M, Cara C, Lauwerys B, Tilt N, Ufuktepe B, Xavier RM, Balsa A, Curtis JR, Mikuls TR, Weinblatt M. Impact of high rheumatoid factor levels on treatment outcomes with certolizumab pegol and adalimumab in patients with rheumatoid arthritis. Rheumatology (Oxford). 2024 Nov 1;63(11):3015-3024. doi: 10.1093/rheumatology/keae435. PMID 39222436
- [Derived] Paul S, Marotte H, Kavanaugh A, Goupille P, Kvien TK, de Longueville M, Mulleman D, Sandborn WJ, Vande Casteele N. Exposure-Response Relationship of Certolizumab Pegol and Achievement of Low Disease Activity and Remission in Patients With Rheumatoid Arthritis. Clin Transl Sci. 2020 Jul;13(4):743-751. doi: 10.1111/cts.12760. Epub 2020 Apr 1. PMID 32100960
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study started to enroll patients in December 2011 and concluded in January 2016.
Pre-assignment Details: Participant Flow refers to the Randomized Treatment Group (RTG) that consisted of all subjects randomized into the study.
Groups:
- CZP+MTX (RTG): Subjects received loading doses of CZP 400mg (200mg/PFS, ie, 2 injections) at Baseline, and Weeks 2 and 4; and CZP 200mg at Weeks 6, 8, and 10.
  Week 12 Responders continued CZP 200mg at Week 12 and every 2 weeks thereafter through Week 102.
  Week 12 Non-Responders were switched to receive ADA 40mg at Week 12 and every 2 weeks through Week 22. At Week 24, Week 12 Non-Responders who did not have DAS28(ESR) LDA or a DAS28(ESR) change from Week 12 reduction of ≥1.2 discontinued ADA treatment and were withdrawn from the Treatment Period.
  All subjects received Methotrexate 15 to 25mg/week orally or subcutaneously from Baseline through Week 104. Regimens could have been changed at Week 52 only. Subjects who could not tolerate these doses could receive MTX at a minimum dose of 10mg/week orally or subcutaneously.
- ADA+MTX (RTG): Subjects received ADA 40mg (40mg/PFS, ie, 1 injection) at Baseline and then every 2 weeks through Week 10. In order to preserve the blind (ie, use of 2 injections) until Week 12, subjects received an injection of PBO in addition to ADA at Baseline, and Weeks 2 and 4.
  Week 12 Responders continued ADA 40mg at Week 12 and every 2 weeks thereafter through Week 102.
  Week 12 Non-Responders were switched to a loading dose of CZP 400mg at Weeks 12, 14, and 16 followed by CZP 200mg every 2 weeks through Week 22. At Week 24, Week 12 Non-Responders who did not have DAS28(ESR) LDA or a DAS28(ESR) change from Week 12 reduction of ≥1.2 discontinued CZP treatment and were withdrawn from the Treatment Period.
  All subjects received Methotrexate 15 to 25mg/week orally or subcutaneously from Baseline through Week 104. Regimens could have been changed at Week 52 only. Subjects who could not tolerate these doses could receive MTX at a minimum dose of 10mg/week orally or subcutaneously.
Period: Week 0 - Week 12
Arm/Group | CZP+MTX (RTG) | ADA+MTX (RTG)
Started | 457 | 458
Completed | 426 | 428
Not Completed | 31 | 30
Not completed — Lack of Efficacy | 0 | 1
Not completed — Protocol Violation | 10 | 16
Not completed — Lost to Follow-up | 1 | 1
Not completed — Withdrawal by Subject | 7 | 2
Not completed — Protocol violation on screening X-ray | 1 | 0
Not completed — Patient decision | 1 | 0
Not completed — Exclusion criteria not met | 1 | 0
Not completed — Investigator decision | 1 | 0
Not completed — Prior history of serious disease | 1 | 0
Not completed — Sponsor decision | 1 | 0
Not completed — Personal reason | 0 | 1
Not completed — Other serious disease | 0 | 1
Not completed — Adverse event (AE), not fatal | 7 | 8
Period: Week 13 - Week 104
Arm/Group | CZP+MTX (RTG) | ADA+MTX (RTG)
Started | 426 | 428
Completed | 287 | 302
Not Completed | 139 | 126
Not completed — Lack of Efficacy | 11 | 12
Not completed — Protocol Violation | 6 | 6
Not completed — Lost to Follow-up | 6 | 5
Not completed — Withdrawal by Subject | 22 | 13
Not completed — Week 24 Non-Responder | 20 | 16
Not completed — Non/bad compliance | 7 | 5
Not completed — Recurrent infections | 1 | 0
Not completed — False positive test | 1 | 2
Not completed — Sponsor request | 4 | 0
Not completed — Withdrawn in error | 1 | 0
Not completed — Exclusion criteria not met | 1 | 0
Not completed — Protocol deviation | 1 | 0
Not completed — Principal investigator retiring | 1 | 0
Not completed — Patient declined Safety Follow Up Visit | 1 | 0
Not completed — Abnormal questionable chest X-ray | 0 | 2
Not completed — Relocation | 0 | 1
Not completed — Sponsor decision | 0 | 2
Not completed — Medical monitor decision | 0 | 2
Not completed — Personal reason | 0 | 1
Not completed — Not completed | 0 | 1
Not completed — Death | 2 | 4
Not completed — Adverse Event | 54 | 54

BASELINE CHARACTERISTICS:
Population: Baseline Characteristics refer to the Randomized Treatment Group (RTG) that consisted of all subjects randomized into the study.
Arm/Group | CZP+MTX (RTG) | ADA+MTX (RTG) | Total Title
Number analyzed (Participants) | 457 | 458 | 915
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 1 | 1
  Between 18 and 65 years | 364 | 372 | 736
  >=65 years | 93 | 85 | 178
Age, Continuous [Mean (Standard Deviation); unit: years]
  Arithmetic mean (standard deviation) | 53.5 (12.3) | 52.9 (12.8) | 53.2 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 360 | 363 | 723
  Male | 97 | 95 | 192

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects Who Met the American College of Rheumatology 20 % (ACR20) Criteria at Week 12
Description: Subjects who met the ACR20 criteria were those subjects with at least 20% improvement from Baseline for Tender Joint Count (TJC), Swollen Joint Count (SJC), and at least 3 of the 5 remaining core set measures: 1) Health Assessment Questionnaire-Disability Index (HAQ-DI), 2) C-reactive Protein (CRP), 3) Patient's Assessment of Arthritis Pain-Visual Analog Scale (PAAP-VAS), 4) Patient's Global Assessment of Disease Activity-Visual Analog Scale (PtGADA-VAS), 5) Physician's Global Assessment of Disease Activity-Visual Analog Scale (PhGA-VAS).
Time Frame: Week 12
Population: The Full Analysis Set (FAS) consisted of all subjects who had a valid Baseline and valid post-Baseline efficacy measurement.
Measure: Number; unit: Percentage of subjects
Groups:
- CZP+MTX (FAS): Subjects received loading doses of CZP 400mg (200mg/PFS, ie, 2 injections) at Baseline, and Weeks 2 and 4; and CZP 200mg at Weeks 6, 8, and 10.
  Week 12 Responders continued CZP 200mg at Week 12 and every 2 weeks thereafter through Week 102.
  Week 12 Non-Responders were switched to receive ADA 40mg at Week 12 and every 2 weeks through Week 22. At Week 24, Week 12 Non-Responders who did not have DAS28(ESR) LDA or a DAS28(ESR) change from Week 12 reduction of ≥1.2 discontinued ADA treatment and were withdrawn from the Treatment Period.
  All subjects received Methotrexate 15 to 25mg/week orally or subcutaneously from Baseline through Week 104. Regimens could have been changed at Week 52 only. Subjects who could not tolerate these doses could receive MTX at a minimum dose of 10mg/week orally or subcutaneously.
- ADA+MTX (FAS): Subjects received ADA 40mg (40mg/PFS, ie, 1 injection) at Baseline and then every 2 weeks through Week 10. In order to preserve the blind (ie, use of 2 injections) until Week 12, subjects received an injection of PBO in addition to ADA at Baseline, and Weeks 2 and 4.
  Week 12 Responders continued ADA 40mg at Week 12 and every 2 weeks thereafter through Week 102.
  Week 12 Non-Responders were switched to a loading dose of CZP 400mg at Weeks 12, 14, and 16 followed by CZP 200mg every 2 weeks through Week 22. At Week 24, Week 12 Non-Responders who did not have DAS28(ESR) LDA or a DAS28(ESR) change from Week 12 reduction of ≥1.2 discontinued CZP treatment and were withdrawn from the Treatment Period.
  All subjects received Methotrexate 15 to 25mg/week orally or subcutaneously from Baseline through Week 104. Regimens could have been changed at Week 52 only. Subjects who could not tolerate these doses could receive MTX at a minimum dose of 10mg/week orally or subcutaneously.
Arm/Group | CZP+MTX (FAS) | ADA+MTX (FAS)
Number analyzed (Participants) | 454 | 454
Percentage of subjects | 69.2 | 71.4
Statistical Analysis 1: Comparison: CZP+MTX (FAS) vs ADA+MTX (FAS); Test type: Superiority or Other; p = 0.467, Regression, Logistic — The odds ratio, CI, and p-value are from a logistic regression model with RTG, gender, Baseline duration of RA (<2 years or >=2 years), and geographic region as factors and age as a covariate; Odds Ratio (OR) = 0.90, 95% CI 2-sided [0.67 to 1.20]

2. Primary Outcome: Percentage of Subjects Who Had a Disease Activity Score 28 [Erythrocyte Sedimentation Rate] (DAS28 [ESR]) ≤ 3.2 at Week 104
Description: DAS28 [ESR] was calculated using the Tender Joint Count (TJC), Swollen Joint Count (SJC), Erythrocyte Sedimentation Rate (ESR in mm/hour), and the Patient's Global Assessment of Disease Activity - Visual Analog Scale (PtGADA-VAS in mm) using the following formula: 0.56 x √ (TJC) + 0.28 x √ (SJC) + 0.70 x lognat (ESR) + 0.014 x Patient Global Assessment of Arthritis, where 28 joints were examined and a lower score indicates less disease activity.
Time Frame: Week 104
Population: as for outcome 1
Measure: Number; unit: Percentage of subjects
Arm/Group | CZP+MTX (FAS) | ADA+MTX (FAS)
Number analyzed (Participants) | 454 | 454
Percentage of subjects | 35.5 | 33.5
Statistical Analysis 1: Comparison: CZP+MTX (FAS) vs ADA+MTX (FAS); Test type: Superiority or Other; p = 0.532, Regression, Logistic — The odds ratio, CI and p-value are from a logistic regression model with RTG, gender, Baseline duration of RA (<2 years or >=2 years), and geographic region as factors and Baseline DAS28(ESR) and age as covariates; Odds Ratio (OR) = 1.09, 95% CI 2-sided [0.82 to 1.45]

3. Secondary Outcome: Percentage of Week 12 Responders Who Had a Disease Activity Score 28 [Erythrocyte Sedimentation Rate] (DAS28 [ESR]) ≤ 3.2 at Week 104
Description: DAS28 [ESR] was calculated using the Tender Joint Count (TJC), Swollen Joint Count (SJC), Erythrocyte Sedimentation Rate (ESR in mm/hour), and the Patient's Global Assessment of Disease Activity - Visual Analog Scale (PtGADA-VAS in mm) using the following formula: 0.56 x √ (TJC) + 0.28 x √ (SJC) + 0.70 x lognat (ESR) + 0.014 x Patient Global Assessment of Arthritis, where 28 joints were examined and a lower score indicates less disease activity.
  The definition of Week 12 responders was DAS28[ESR] Low Disease Activity (LDA) (ie ≤ 3.2) or an improvement of ≥ 1.2 in DAS28[ESR] relative to Baseline.
Time Frame: Week 104
Population: Week 12 Responders were defined as those with DAS28(ESR) LDA (defined as DAS28[ESR] ≤3.2) or a DAS28(ESR) CFB reduction of ≥1.2 at Week 12.
Measure: Number; unit: Percentage of subjects
Groups:
- CZP+MTX (Week 12 Responder Set): CZP 400 mg at Baseline, Week 2 and Week 4, followed by a maintenance dose of 200 mg every 2 Weeks until Week 102.
  All subjects received Methotrexate 15 to 25mg/week orally or subcutaneously from Baseline through Week 104. Regimens could have been changed at Week 52 only. Subjects who could not tolerate these doses could receive MTX at a minimum dose of 10mg/week orally or subcutaneously.
- ADA+MTX (Week 12 Responder Set): ADA 40 mg at Baseline and then every 2 Weeks until Week 102. Subjects received PBO in addition to ADA at baseline and weeks 2 and 4 in order to maintain the blinding.
  All subjects received Methotrexate 15 to 25mg/week orally or subcutaneously from Baseline through Week 104. Regimens could have been changed at Week 52 only. Subjects who could not tolerate these doses could receive MTX at a minimum dose of 10mg/week orally or subcutaneously.
Arm/Group | CZP+MTX (Week 12 Responder Set) | ADA+MTX (Week 12 Responder Set)
Number analyzed (Participants) | 353 | 361
Percentage of subjects | 45.6 | 42.4

4. Secondary Outcome: Percentage of Subjects Who Met the American College of Rheumatology 20 % (ACR20) Criteria at Week 6
Description: as for outcome 1
Time Frame: Week 6
Population: as for outcome 1
Measure: Number; unit: Percentage of subjects
Arm/Group | CZP+MTX (FAS) | ADA+MTX (FAS)
Number analyzed (Participants) | 454 | 454
Percentage of subjects | 64.5 | 60.8

5. Secondary Outcome: Percentage of Subjects Who Had a Disease Activity Score 28 [Erythrocyte Sedimentation Rate] (DAS28 [ESR]) ≤ 3.2 at Week 6
Description: as for outcome 2
Time Frame: Week 6
Population: as for outcome 1
Measure: Number; unit: Percentage of subjects
Arm/Group | CZP+MTX (FAS) | ADA+MTX (FAS)
Number analyzed (Participants) | 454 | 454
Percentage of subjects | 20.5 | 18.1

6. Secondary Outcome: Percentage of Subjects Who Had a Disease Activity Score 28 [Erythrocyte Sedimentation Rate] (DAS28 [ESR]) ≤ 3.2 at Week 12
Description: as for outcome 2
Time Frame: Week 12
Population: as for outcome 1
Measure: Number; unit: Percentage of subjects
Arm/Group | CZP+MTX (FAS) | ADA+MTX (FAS)
Number analyzed (Participants) | 454 | 454
Percentage of subjects | 30.4 | 29.7

7. Secondary Outcome: Percentage of Subjects With a Disease Activity Score 28 [Erythrocyte Sedimentation Rate] (DAS28 [ESR]) ≤ 3.2 at Week 104, in Subjects Responding at Both Week 6 and Week 12
Description: DAS28 [ESR] was calculated using the Tender Joint Count (TJC), Swollen Joint Count (SJC), Erythrocyte Sedimentation Rate (ESR in mm/hour), and the Patient's Global Assessment of Disease Activity - Visual Analog Scale (PtGADA-VAS in mm) using the following formula: 0.56 x √ (TJC) + 0.28 x √ (SJC) + 0.70 x lognat (ESR) + 0.014 x Patient Global Assessment of Arthritis, where 28 joints were examined and a lower score indicates less disease activity.
  The definition of Week 6/12 responders was DAS28[ESR] Low Disease Activity (LDA) (ie ≤ 3.2) or an improvement of ≥ 1.2 in DAS28[ESR] relative to Baseline.
Time Frame: Week 104
Population: Week 12 Responders were defined as those with DAS28(ESR) LDA (defined as DAS28[ESR] ≤3.2) or a DAS28(ESR) CFB reduction of ≥1.2 at Week 12. Only subjects responding at both Week 6 and Week 12 are included in this analysis.
Measure: Number; unit: Percentage of subjects
Arm/Group | CZP+MTX (Week 12 Responder Set) | ADA+MTX (Week 12 Responder Set)
Number analyzed (Participants) | 310 | 298
Percentage of subjects | 47.7 | 46.6

8. Secondary Outcome: Change From Baseline in the Health Assessment Questionnaire-Disability Index (HAQ-DI) at Week 104
Description: HAQ-DI was derived based on the mean of individual scores in 8 categories of daily living actives (using 20 questions). Each question was scored 0-3 (0 = without any difficulty, 1 = with some difficulty, 2 = with much difficulty, and 3 = unable to do), and the total HAQ-DI was scored on the scale of 0-3 as well. Change from Baseline was computed as the value at Week 104 minus the Baseline value. A negative value in Change from Baseline indicates an improvement.
Time Frame: From Baseline to Week 104
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Units on a Scale
Arm/Group | CZP+MTX (FAS) | ADA+MTX (FAS)
Number analyzed (Participants) | 454 | 454
Units on a Scale | -0.62 (0.03) | -0.72 (0.03)

9. Secondary Outcome: Kaplan-Meier Estimates of Proportion of Subjects Who Discontinued After Response at Week 12
Description: Response at Week 12 means that a subject had either a Disease Activity Score 28 [Erythrocyte Sedimentation Rate] (DAS28 [ESR]) ≤ 3.2 at Week 12 or had a reduction of DAS28 [ESR] ≥ 1.2 from Baseline to Week 12. Kaplan-Meier Estimates of Proportion of Subjects Discontinued are presented per study week (days relative to Week 12 visit).
Time Frame: From Week 12 up to Week 104
Population: as for outcome 3
Measure: Number; unit: proportion of subjects
Arm/Group | CZP+MTX (Week 12 Responder Set) | ADA+MTX (Week 12 Responder Set)
Number analyzed (Participants) | 353 | 361
proportion of subjects
  Week 13 (Day 7) | 0 | 0.0028
  Week 26 (Day 98) | 0.0198 | 0.0332
  Week 39 (Day 189) | 0.0453 | 0.0609
  Week 52 (Day 280) | 0.0963 | 0.0886
  Week 65 (Day 371) | 0.1643 | 0.1607
  Week 78 (Day 462) | 0.2181 | 0.1967
  Week 91 (Day 553) | 0.2408 | 0.2105
  Week 104 (Day 644) | 0.2635 | 0.2247

ADVERSE EVENTS:
Time Frame: During the entire study period (From Week -4 to Week 104).
Description: The AEs of subjects who switched study treatment at Week 12 (W12) were presented under the original treatment group if they occurred after the 1st administration of study treatment (W0) until the day before W12 treatment administration, and were presented under the switched treatment group if they occurred after the W12 treatment administration up to and including 70 days after the last injection. Subjects who switched treatment at W12 were included in both CZP+MTX(SS) and ADA+MTX(SS) group.
Groups:
- CZP+MTX (SS): All subjects who received at least 1 dose of Certolizumab pegol (CZP). All adverse events that occurred when the subject was receiving CZP treatment are summarized in this group.
- ADA+MTX (SS): All subjects who received at least 1 dose of Adalimumab (ADA). All adverse events that occurred when the subject was receiving ADA treatment are summarized in this group.
Arm/Group | CZP+MTX (SS) | ADA+MTX (SS)
Serious Adverse Events (participants affected / at risk) | 67/516 | 58/523
Other Adverse Events (participants affected / at risk) | 269/516 | 244/523
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CZP+MTX (SS) (N=516) | ADA+MTX (SS) (N=523)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Aortic valve incompetence (Cardiac disorders) | 0 (0) | 1 (1)
Aortic valve stenosis (Cardiac disorders) | 0 (0) | 1 (1)
Stress cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 2 (2) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 1 (1)
Cardiogenic shock (Cardiac disorders) | 0 (0) | 1 (1)
Angina unstable (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1) | 1 (1)
Ophthalmic vein thrombosis (Eye disorders) | 0 (0) | 1 (1)
Diplopia (Eye disorders) | 1 (1) | 0 (0)
Obstruction gastric (Gastrointestinal disorders) | 1 (1) | 0 (0)
Chronic gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1)
Irritable bowel syndrome (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal stenosis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Anorectal varices (Gastrointestinal disorders) | 1 (1) | 0 (0)
Sudden death (General disorders) | 0 (0) | 1 (1)
Impaired healing (General disorders) | 1 (1) | 0 (0)
Systemic inflammatory response syndrome (General disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 2 (2)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 4 (4)
Hepatotoxicity (Hepatobiliary disorders) | 1 (1) | 0 (0)
Drug-induced liver injury (Hepatobiliary disorders) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Appendicitis perforated (Infections and infestations) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 1 (1)
Perirectal abscess (Infections and infestations) | 1 (1) | 0 (0)
Bronchopulmonary aspergillosis (Infections and infestations) | 0 (0) | 1 (1)
Mycobacterial infection (Infections and infestations) | 2 (2) | 0 (0)
Bronchitis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 2 (2)
Clostridium difficile infection (Infections and infestations) | 1 (1) | 0 (0)
Oophoritis (Infections and infestations) | 1 (1) | 0 (0)
Hepatitis A (Infections and infestations) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1)
Pneumonia (Infections and infestations) | 6 (6) | 5 (5)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Subcutaneous abscess (Infections and infestations) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 1 (1)
Disseminated tuberculosis (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 2 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (2) | 1 (1)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 0 (0) | 1 (1)
Joint injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Subdural heamatoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Lower limb fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ancle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Bone disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Invertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Torticollis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Tendon disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Borderline mucinous tumour of ovary (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Ovarian adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cerebral haematoma (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral ischaemia (Nervous system disorders) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Coma (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Generalised tonic-clonic seizure (Nervous system disorders) | 1 (1) | 0 (0)
Amnesia (Nervous system disorders) | 1 (1) | 0 (0)
Post herpetic neuralgia (Nervous system disorders) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0)
Abortion (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Pregnancy with contraceptive device (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Adjustment disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Anxiety disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Bipolar disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1)
Cervical dysplasia (Reproductive system and breast disorders) | 0 (0) | 2 (2)
Menorrhagia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Osteosynthesis (Surgical and medical procedures) | 1 (1) | 0 (0)
Hip arthroplasty (Surgical and medical procedures) | 0 (0) | 1 (1)
Venous thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Peripheral venous disease (Vascular disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Venous thrombosis limb (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CZP+MTX (SS) (N=516) | ADA+MTX (SS) (N=523)
Diarrhoea (Gastrointestinal disorders) | 31 (36) | 23 (26)
Nasopharyngitis (Infections and infestations) | 79 (116) | 67 (106)
Upper respiratory tract infection (Infections and infestations) | 53 (74) | 60 (80)
Urinary tract infection (Infections and infestations) | 43 (58) | 51 (65)
Latent tuberculosis (Infections and infestations) | 31 (31) | 27 (27)
Sinusitis (Infections and infestations) | 31 (35) | 21 (31)
Bronchitis (Infections and infestations) | 29 (33) | 25 (26)
Headache (Nervous system disorders) | 55 (62) | 47 (77)
Cough (Respiratory, thoracic and mediastinal disorders) | 21 (26) | 28 (35)
Hypertension (Vascular disorders) | 37 (42) | 31 (34)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days